CLINICAL TRIAL: NCT02688530
Title: Intravenous Dexamethasone for Prolongation of Analgesia Following Supraclavicular Brachial Plexus Block for Shoulder Arthroscopy: A Randomized, Controlled, Phase IV Dose-Response Study
Brief Title: Intravenous Dexamethasone on Supraclavicular Brachial Plexus Block for Shoulder Arthroscopy
Acronym: SCB & IV Dex
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 2015-853
Record Dates: First submitted 2016-02-18; First posted 2016-02-23 (Estimated); Results first posted 2022-05-13 (Actual); Last update posted 2022-05-13 (Actual); Status verified 2022-05

CONDITIONS: Shoulder Arthroscopy; Pain
MeSH Terms: conditions — Pain | interventions — Sodium Chloride; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- 0mg IV Dexamethasone (Placebo Comparator): 0mg IV Dexamethasone
  Interventions: Drug: IV Saline
- 4mg IV Dexamethasone (Experimental): 4mg IV Dexamethasone
  Interventions: Drug: IV Dexamethasone 4mg
- 6mg IV Dexamethasone (Experimental): 6mg IV Dexamethasone
  Interventions: Drug: IV Dexamethasone 6mg
- 8mg IV Dexamethasone (Experimental): 8mg IV Dexamethasone
  Interventions: Drug: IV Dexamethasone 8mg

INTERVENTIONS:
Drug: IV Saline
  Arms: 0mg IV Dexamethasone
Drug: IV Dexamethasone 4mg
  Arms: 4mg IV Dexamethasone
Drug: IV Dexamethasone 6mg
  Arms: 6mg IV Dexamethasone
Drug: IV Dexamethasone 8mg
  Arms: 8mg IV Dexamethasone

SUMMARY:
Previous studies have confirmed that IV dexamethasone prolongs brachial plexus blocks. However, these studies only used fixed doses of IV dexamethasone at relatively high doses, which could potentially lead to increased glucose levels, delayed wound healing, and unintended side effects. There remains a paucity of research on the effective dose range of IV dexamethasone for the prolongation of supraclavicular blocks. The optimal dosage of IV dexamethasone for prolongation of analgesia vs. motor block prolongation from supraclavicular blocks in shoulder surgery has yet to be delineated.

DETAILED DESCRIPTION:
Numerous studies have confirmed that perineural dexamethasone prolongs bupivacaine and ropivacaine brachial plexus blocks by approximately 10 hours (from approx. 12 to 22 hours) without clinical evidence of toxicity. However, perineural toxicity in an animal model has raised concern about its use as a peripheral nerve block adjuvant. Moreover, recent studies suggest that high dose IV dexamethasone (810mg) prolongs analgesia to a similar degree as perineural dexamethasone for interscalene, supraclavicular and sciatic nerve blocks performed with ropivacaine and bupivacaine. However these studies only utilized fixed, high level doses of IV dexamethasone. Moreover, there remains a concern that high dose IV dexamethasone may lead to postoperative hyperglycemia and could possibly increase the risk of postoperative wound infection. Open surgery under general anesthesia has been shown to increase blood glucose levels with a peak at approximately 2 hours post-induction and results have been conflicting regarding whether or not IV dexamethasone causes greater increase. To the investigators' knowledge, it is not yet known if arthroscopic surgery under regional anesthesia triggers a similar increase in blood glucose levels and if this is impacted by administration of IV dexamethasone. The investigators aim to identify the duration of supraclavicular block prolongation that can be expected over a range of doses of IV dexamethasone. The investigators also seek to identify what association, if any, is noted between IV dexamethasone and changes in blood glucose levels after shoulder surgery with regional anesthesia and sedation. Finally, the investigators will collect data on side effects and postoperative complications, if any, in patients receiving a range of doses of IV dexamethasone.

ELIGIBILITY:
Inclusion Criteria:

- Patients undergoing shoulder arthroscopy under regional anesthesia

Exclusion Criteria:

* General anesthesia
* Contraindication to regional anesthesia
* Pre-existing neuropathy in the surgical limb
* Diabetes Mellitus
* History of postoperative nausea and vomiting &/ or motion sickness
* Procedures involving biceps tenotomy
* Peri-articular cocktail injections given intraoperatively to augment pain relief
* Chronic pain (daily opioid and/or gabapentinoid use for 6 weeks)
* Open surgical procedures
* Corticosteroid injection within 1 month
* Patients on systemic oral or IV steroid therapy within 6 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2016-05; Primary Completion 2017-11-19 (Actual); Study Completion 2017-11-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Meghan Kirksey, MD, PhD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- 0mg IV Dexamethasone: 0mg IV Dexamethasone
  IV Saline
- 4mg IV Dexamethasone: 4mg IV Dexamethasone
  IV Dexamethasone 4mg
- 6mg IV Dexamethasone: 6mg IV Dexamethasone
  IV Dexamethasone 6mg
- 8mg IV Dexamethasone: 8mg IV Dexamethasone
  IV Dexamethasone 8mg
Period: Overall Study
Arm/Group | 0mg IV Dexamethasone | 4mg IV Dexamethasone | 6mg IV Dexamethasone | 8mg IV Dexamethasone
Started | 35 | 35 | 35 | 35
Completed | 35 | 34 | 33 | 35
Not Completed | 0 | 1 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 0mg IV Dexamethasone | 4mg IV Dexamethasone | 6mg IV Dexamethasone | 8mg IV Dexamethasone | Total
Number analyzed (Participants) | 35 | 34 | 33 | 35 | 137
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 28 | 27 | 25 | 32 | 112
  >=65 years | 7 | 7 | 8 | 3 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] — full range
  years | 49 (16) | 50 (17) | 52 (15) | 49 (12) | 50 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 6 | 10 | 10 | 42
  Male | 19 | 28 | 23 | 25 | 95
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 1 | 0 | 0 | 1 | 2
  Race: Black/African American | 1 | 1 | 1 | 0 | 3
  Race: White | 33 | 32 | 32 | 32 | 129
  Race: Unknown | 0 | 1 | 0 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 35 | 34 | 33 | 35 | 137

OUTCOME MEASURES:

1. Primary Outcome: Duration of Analgesia From a Supraclavicular Block Performed for Shoulder Arthroscopy
Description: Defined as time from block placement until "pain relief from the block completely wears off" in the operative shoulder.
Time Frame: Day of Surgery until Post-Operative Day 3 (if the block persists)
Measure: Median (95% Confidence Interval); unit: Hours
Arm/Group | 0mg IV Dexamethasone | 4mg IV Dexamethasone | 6mg IV Dexamethasone | 8mg IV Dexamethasone
Number analyzed (Participants) | 35 | 34 | 33 | 35
Hours | 17.4 [12 to 23.4] | 22.7 [18.1 to 28.1] | 20.2 [17.5 to 25] | 19.8 [16.5 to 24.5]

2. Secondary Outcome: Duration of Motor Block From the Supraclavicular Block
Description: Defined as the time from block placement to restoration of normal strength at both the wrist and elbow.
Time Frame: Day of Surgery until Post-Operative Day 3 (if the block persists)
Population: shoulder arthroscopy
Measure: Median (95% Confidence Interval); unit: Hours
Arm/Group | 0mg IV Dexamethasone | 4mg IV Dexamethasone | 6mg IV Dexamethasone | 8mg IV Dexamethasone
Number analyzed (Participants) | 35 | 34 | 33 | 35
Hours | 10.5 [8.3 to 14.9] | 19.7 [14.8 to 21.9] | 18.3 [15 to 21.4] | 14.7 [12.7 to 18.7]

3. Secondary Outcome: Blood Glucose Levels
Description: Fingerstick blood glucose test to be administered before and 1-hour and 2-hours after IV dexamethasone administration.
Time Frame: Day of Surgery - before and 1-hour and 2-hours after IV Dexamethasone administration
Population: Prior to IV Dexamethasone, 1-hour and 2-hours after IV Dexamethasone administration
Measure: Median (Standard Deviation); unit: mg/dL
Arm/Group | 0mg IV Dexamethasone | 4mg IV Dexamethasone | 6mg IV Dexamethasone | 8mg IV Dexamethasone
Number analyzed (Participants) | 35 | 34 | 31 | 33
mg/dL
  Prior to IV Dexamethasone | 102 (15) | 108 (14) | 104 (16) | 105 (18)
  1 hour after IV Dexamethasone | 119 (14) | 122 (17) | 119 (18) | 126 (18)
  2 hours after IV Dexamethasone | 102 (20) | 125 (31) | 110 (23) | 110 (27)

4. Secondary Outcome: Occurrence of Postoperative Neuropraxia
Description: Documentation of any of these occurrences will be obtained from the surgeons and/or medical charts after the postoperative follow up visit.
Time Frame: Post-Operative Day 21
Measure: Count of Participants; unit: Participants
Arm/Group | 0mg IV Dexamethasone | 4mg IV Dexamethasone | 6mg IV Dexamethasone | 8mg IV Dexamethasone
Number analyzed (Participants) | 28 | 29 | 27 | 28
Participants | 0 | 1 | 0 | 0

5. Secondary Outcome: Occurrence of Postoperative Wound Infection
Description: as for outcome 4
Time Frame: Post-Operative Day 21
Measure: Count of Participants; unit: Participants
Arm/Group | 0mg IV Dexamethasone | 4mg IV Dexamethasone | 6mg IV Dexamethasone | 8mg IV Dexamethasone
Number analyzed (Participants) | 28 | 29 | 27 | 28
Participants | 0 | 0 | 0 | 0

6. Secondary Outcome: Average Daily Pain Scores at Rest and With Movement
Description: Using the Numeric Rating Scale (NRS) Pain obtained by patient interview. Lower numbers represent less pain and better outcomes. The scale range is from 0 (no pain) to 10 (worst pain possible).
Time Frame: Day of Surgery until Post-Operative Day 3 (if the block persists)
Population: Average daily pain scores Pre-Op to POD3 at rest and with movement.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0mg IV Dexamethasone | 4mg IV Dexamethasone | 6mg IV Dexamethasone | 8mg IV Dexamethasone
Number analyzed (Participants) | 35 | 34 | 33 | 35
score on a scale
  Pre-Op Average Pain Score at rest | 2.6 (1.9) | 3 (2.5) | 2.4 (2.4) | 2.5 (2.5)
  POD0 Average Pain Score at rest: number analyzed (Participants) | 35 | 34 | 32 | 35
  POD0 Average Pain Score at rest | 0.4 (1.1) | 0.2 (0.7) | 0.4 (0.9) | 0.5 (1.6)
  POD1 Average Pain Score at rest: number analyzed (Participants) | 35 | 33 | 33 | 35
  POD1 Average Pain Score at rest | 4.1 (2.5) | 3.2 (2.1) | 3.1 (2.8) | 3 (2.5)
  POD2 Average Pain Score at rest: number analyzed (Participants) | 33 | 34 | 30 | 33
  POD2 Average Pain Score at rest | 2.9 (2.1) | 3.7 (1.8) | 3.3 (2.7) | 3.1 (2.4)
  POD3 Average Pain Score at rest: number analyzed (Participants) | 2 | 3 | 1 | 3
  POD3 Average Pain Score at rest | 0.5 (0.7) | 4 (1.7) | 3 (0) | 2 (2)
  Pre-Op Average Pain Score with Movement | 4.6 (2.3) | 4.8 (2.3) | 4.6 (2.4) | 4.7 (2.7)
  POD0 Average Pain Score with Movement: number analyzed (Participants) | 19 | 19 | 17 | 17
  POD0 Average Pain Score with Movement | 0.5 (1.4) | 0.3 (0.8) | 0.2 (0.5) | 0.4 (1.7)
  POD1 Average Pain Score with Movement: number analyzed (Participants) | 35 | 33 | 33 | 35
  POD1 Average Pain Score with Movement | 5.2 (2.6) | 4.7 (2.2) | 4.8 (3.1) | 4.2 (3.3)
  POD2 Average Pain Score with Movement: number analyzed (Participants) | 33 | 34 | 30 | 33
  POD2 Average Pain Score with Movement | 4.6 (2.6) | 5.1 (2.3) | 5 (2.3) | 4.8 (2.3)
  POD3 Average Pain Score with Movement: number analyzed (Participants) | 2 | 3 | 1 | 3
  POD3 Average Pain Score with Movement | 6 (2.8) | 5 (3) | 6 (0) | 1.7 (1.5)

7. Secondary Outcome: Worst Daily Pain Scores at Rest and With Movement
Description: Using the numeric pain rating scale (NRS), will be obtained by patient interview. Lower numbers represent less pain and better outcomes. The scale range is from 0 (no pain) to 10 (worst pain possible).
Time Frame: Day of Surgery until Post-Operative Day 3 (if the block persists)
Population: Worst Daily Pain Scores at rest and with movement from Pre-Op to POD3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0mg IV Dexamethasone | 4mg IV Dexamethasone | 6mg IV Dexamethasone | 8mg IV Dexamethasone
Number analyzed (Participants) | 35 | 34 | 33 | 35
score on a scale
  Pre-Op Worst Pain Score at rest | 3.4 (2.1) | 3.3 (2.9) | 3.4 (2.6) | 3.6 (3.1)
  POD0 Worst Pain Score at rest: number analyzed (Participants) | 35 | 34 | 32 | 35
  POD0 Worst Pain Score at rest | 0.6 (1.5) | 0.2 (0.7) | 0.5 (1.3) | 1.1 (2.7)
  POD1 Worst Pain Score at rest: number analyzed (Participants) | 35 | 33 | 33 | 35
  POD1 Worst Pain Score at rest | 6.3 (2.9) | 4.6 (2.8) | 5.4 (3.2) | 5.1 (3.5)
  POD2 Worst Pain Score at rest: number analyzed (Participants) | 33 | 34 | 30 | 33
  POD2 Worst Pain Score at rest | 4.7 (3) | 5.4 (2.3) | 5.1 (2.8) | 4.5 (3.3)
  POD3 Worst Pain Score at rest: number analyzed (Participants) | 2 | 3 | 1 | 3
  POD3 Worst Pain Score at rest | 2 (1.4) | 6.3 (2.9) | 5 (0) | 4.3 (3.5)
  Pre-Op Worst Pain Score with Movement | 6.1 (2.7) | 6.5 (2.4) | 6.4 (2.5) | 6.9 (2.7)
  POD0 Worst Pain Score with Movement: number analyzed (Participants) | 19 | 19 | 17 | 17
  POD0 Worst Pain Score with Movement | 0.6 (1.9) | 0.3 (0.8) | 0.3 (0.8) | 1.2 (3.3)
  POD1 Worst Pain Score with Movement: number analyzed (Participants) | 35 | 33 | 33 | 35
  POD1 Worst Pain Score with Movement | 7.3 (2.6) | 5.9 (2.7) | 6.5 (3.1) | 5.7 (3.4)
  POD2 Worst Pain Score with Movement: number analyzed (Participants) | 33 | 34 | 30 | 33
  POD2 Worst Pain Score with Movement | 6.5 (2.9) | 6.8 (2.2) | 6.7 (2.2) | 6.3 (2.5)
  POD3 Worst Pain Score with Movement: number analyzed (Participants) | 2 | 3 | 1 | 3
  POD3 Worst Pain Score with Movement | 7 (1.4) | 6.7 (3.2) | 7 (0) | 3.7 (3.2)

8. Secondary Outcome: Patient Satisfaction With Postoperative Analgesia
Description: Patient satisfaction with postoperative analgesia will be obtained by patient interview. Lower numbers represent worse outcomes. The scale range is from 0 (worst) to 10 (best).
Time Frame: Post-Operative Day 2 or Post-Operative Day 3 (if the block persists)
Population: Patient Satisfaction with Post-Op Analgesia
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0mg IV Dexamethasone | 4mg IV Dexamethasone | 6mg IV Dexamethasone | 8mg IV Dexamethasone
Number analyzed (Participants) | 28 | 29 | 27 | 28
score on a scale | 9.1 (1.2) | 8.9 (1.6) | 9.2 (1.2) | 8.7 (1.7)

9. Secondary Outcome: Cumulative Daily Opioid Usage
Description: Dosages (reported in Morphine equivalent units) of opioid medication obtained by medical records and/or by patient interview.
Time Frame: Recovery Room until Post-Operative Day 3 (if block persists)
Population: Cumulative Daily Opioid Usage
Measure: Mean (Standard Deviation); unit: oral morphine equivalent units (mg)
Arm/Group | 0mg IV Dexamethasone | 4mg IV Dexamethasone | 6mg IV Dexamethasone | 8mg IV Dexamethasone
Number analyzed (Participants) | 35 | 34 | 33 | 35
oral morphine equivalent units (mg)
  POD 1 (0-24hrs) | 31 (23.7) | 30.5 (29.3) | 30.7 (25.9) | 31.3 (34.1)
  POD2 (24-48hrs): number analyzed (Participants) | 34 | 34 | 32 | 34
  POD2 (24-48hrs) | 22.3 (28.2) | 27.4 (41.4) | 32.6 (29.3) | 36.5 (47.5)

ADVERSE EVENTS:
Time Frame: These protocol deviations were between 4/7/17-10/9/2017. Patients were followed for 3 days after surgery.
Groups:
- 0mg IV Dexamethasone: 0 mg IV Dexamethasone Adverse Event
- 4mg IV Dexamethasone: 4 mg IV Dexamethasone Adverse Event
- 6mg IV Dexamethasone: 6 mg IV Dexamethasone Adverse Event
- 8mg IV Dexamethasone: 8 mg IV Dexamethasone Adverse Event
Arm/Group | 0mg IV Dexamethasone | 4mg IV Dexamethasone | 6mg IV Dexamethasone | 8mg IV Dexamethasone
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/34 | 0/33 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/34 | 0/33 | 0/35
Other Adverse Events (participants affected / at risk) | 4/35 | 2/34 | 6/33 | 3/35
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0mg IV Dexamethasone (N=35) | 4mg IV Dexamethasone (N=34) | 6mg IV Dexamethasone (N=33) | 8mg IV Dexamethasone (N=35)
Protocol Deviation (Surgical and medical procedures) | 4 (4) | 2 (2) | 6 (6) | 3 (3) — Medication dosage changes, change of procedure during surgery. These were reported as protocol deviations

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-29): https://cdn.clinicaltrials.gov/large-docs/30/NCT02688530/Prot_SAP_000.pdf